CLINICAL TRIAL: NCT02342249
Title: A Phase 2b, Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter Study of 2 Dose Levels of VX 787 Administered as Monotherapy and One Dose Level of VX-787 Administered in Combination With Oseltamivir for the Treatment of Acute Uncomplicated Seasonal Influenza A in Adult Subjects
Brief Title: Study of Acute Uncomplicated Seasonal Influenza A in Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR107745; VX-787FLZ2001 (Other: Janssen Research & Development, LLC); VX14-787-103 (Other: Janssen Research & Development, LLC); 2014-004068-39 (EudraCT Number)
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Influenza A
Keywords: Influenza A
MeSH Terms: interventions — pimodivir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VX-787 Placebo BID + Oseltamivir Placebo BID (Placebo Comparator): Subjects will receive 10 doses of matching placebo of VX-787 and Oseltamivir twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5-6 days.
  Interventions: Drug: Placebo
- VX-787 300 mg BID + Oseltamivir Placebo BID (Active Comparator): Subjects will receive 10 doses of VX-787 300 milligram (mg) tablet along with matching placebo of Oseltamivir twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5-6 days.
  Interventions: Drug: VX-787 300 mg; Drug: Placebo
- VX-787 600 mg BID + Oseltamivir Placebo BID (Active Comparator): Subjects will receive 10 doses of VX-787 600 mg (2*300 mg tablets) along with matching placebo of Oseltamivir twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5-6 days.
  Interventions: Drug: VX-787 600 mg; Drug: Placebo
- VX-787 600 mg BID + Oseltamivir 75 mg BID (Active Comparator): Subjects will receive 10 doses of VX-787 600 mg tablets (2*300 mg tablets) along with 75 mg Oseltamivir capsule twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5-6 days.
  Interventions: Drug: VX-787 600 mg; Drug: Oseltamivir 75 mg

INTERVENTIONS:
Drug: VX-787 300 mg — A oral dose of 300 mg VX-787 tablet will be administered over 5-6 days.
  Other Names: JNJ-63623872
  Arms: VX-787 300 mg BID + Oseltamivir Placebo BID
Drug: VX-787 600 mg — A oral dose of VX-787 600 mg (formulated as 2*300 mg tablets) will be administered over 5-6 days.
  Other Names: JNJ-63623872
  Arms: VX-787 600 mg BID + Oseltamivir 75 mg BID; VX-787 600 mg BID + Oseltamivir Placebo BID
Drug: Oseltamivir 75 mg — A oral dose of 75 mg Oseltamivir capsule will be administered over 5-6 days.
  Arms: VX-787 600 mg BID + Oseltamivir 75 mg BID
Drug: Placebo — Subjects will receive matching placebo of Oseltamivir
  Arms: VX-787 300 mg BID + Oseltamivir Placebo BID; VX-787 600 mg BID + Oseltamivir Placebo BID; VX-787 Placebo BID + Oseltamivir Placebo BID

SUMMARY:
The purpose of this study is to evaluate the antiviral effect, as measured by viral titer in nasal secretions in adults with acute uncomplicated seasonal influenza A following administration of VX-787.

ELIGIBILITY:
Inclusion Criteria: Part A

1. Willing and able to comply with the NP swab procedure
2. Subject will sign and date an informed consent form (ICF)
3. Presenting to the clinic with symptoms suggestive of a diagnosis of acute influenza. Symptoms include oral temperature ≥38°C (100.4°F) within the prior 24 hours, at least 1 respiratory symptom AND at least 1 systemic symptom.
4. Understand that no study treatment will be provided to subjects in Part A but that they are free to receive any treatment considered appropriate by their physician

Part B

1. Willing and able to comply with study requirements including treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures
2. Subject will sign and date an ICF
3. Present to the clinic with symptoms suggestive of a diagnosis of acute influenza. Symptoms include documented oral temperature ≥38°C (100.4°F) any time during the screening process, at least 1 respiratory symptom AND at least 1 systemic symptom, both scored as at least "moderate".
4. The time of onset of flu-like symptoms to the time anticipated for the start of treatment must be ≤48 hours. Onset of symptoms is defined as the first time (within 1 hour) the subject becomes aware of respiratory or systemic symptoms compatible with the flu or experiences an oral temperature ≥38°C (100.4°F)
5. Positive Rapid Influenza Diagnostic Test for influenza type A
6. Body mass index (BMI) of 18.0 to 33.0 kg/m2, inclusive, and a total body weight >50 kg

Exclusion Criteria: Part B

1. History of any illness or any clinical condition that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject.
2. Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy, or other gastrointestinal tract surgery, except appendectomy).
3. Immunized (intranasal or injected vaccine) against influenza in the 6 months before study entry.
4. At Screening, an ECG that is abnormal and deemed by the investigator(s) to be clinically significant.
5. For female subjects: Pregnant or nursing subjects and female subjects of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol.
6. For male subjects, unwilling to comply with contraception requirements as outlined in the study protocol.
7. Blood donation (of approximately 1 pint [500 mL] or more) within 56 days before the first study drug dose.
8. Use of the following medications:

   * Influenza antiviral medication (oseltamivir, zanamivir, rimantidine, or amantadine) within 14 days or ribavirin within 6 months of screening.
   * Substrates of OATP1B1 and/or OATP1B3, including atrasentan, bosentan, ezetimibe, glyburide, irinotecan, repaglinide, rifampin, telmisartan, valsartan, and olmesartan, from Day 1 through the last dose of study drug. "Statins" (i.e., HMG CoA reductase inhibitors) may be continued, but subjects should be cautioned and observed for potential "statin"-related toxicity. Alternatively, subjects can abstain from statins for the duration of study drug dosing.
   * Strong inhibitors or inducers of CYP3A metabolism, including carbamazepine, clarithromycin, HIV and HCV protease inhibitors, itraconazole, ketoconazole, nefazodone, phenytoin, posaconazole, rifampin, St. John's wort, telithromycin, and voriconazole from 2 weeks prior to the first dose of study drug until the last PK sample is collected on Day 8.
   * An investigational drug or device 30 days before the first dose of study drug, 5 half lives before the first dose of study drug, or time determined by local requirements, whichever is longest.
9. History of excessive alcohol consumption.
10. History of known or current usage of drugs of abuse.
11. Hospitalized subjects and subjects with bacterial infections requiring systemic antibacterial agents at the time of screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the log10 Nasal Viral Load on Day 8 | Day 8
  Area under the curve (AUC) of the log10 nasal viral load is measured by quantitative reverse transcriptase polymerase chain reaction (qRT-PCR).

SECONDARY OUTCOMES:
Time to Resolution of Influenza Symptoms After Initiation of Study Drug | Baseline up to Day 14
  Estimated acceleration factors expressed as the ratio of the time to resolution of influenza symptoms as compared to placebo time to negativity. Resolution of influenza symptoms was the time of the first of 3 evaluations (over 24 hours) in which all symptom scores for each of the 3 assessments are 0 or 1 for all 7 primary influenza symptoms (cough, sore throat, headache, nasal stuffiness, feverishness or chills, muscle or joint pain, and fatigue) of the Flu-iiQ^TM. The Flu-iiQ^TM questionnaire consists of 4 modules, including 1 module assessing influenza symptoms, 1 module assessing the impact of influenza on normal functioning, and 2 modules assessing the impact of influenza on the subject's emotional state. The Influenza Symptom assessment (Module 1) is scored on a 4 point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe) for each of 10 influenza symptoms.
Safety and tolerability based on assessment of adverse events, clinical laboratory assessments, 12-lead electrocardiograms (ECGs), and vital signs | Day 14
Antiviral effect and viral kinetics composite | Days 1 - 8
  Antiviral effect and viral kinetics in relation to:
  * Duration of viral shedding in nasal secretions by qRT-PCR and viral culture
  * AUC of the log10 viral load measured by viral culture
  * Peak viral shedding titer by qRT-PCR and viral culture.
Clinical composite symptom scores | Day 14
  Clinical symptom scores
  * Composite symptom score AUC
  * Time to peak of composite symptom score,
  * Duration and time to resolution of composite symptom score from peak
Pharmacokinetic parameters of VX787, as determined by population analysis | Day 14
  A population Pharmacokinetic Pharmacodynamic analysis of plasma concentration data of VX-787 will be performed using the nonlinear mixed effects modeling approach.
Viral sequence analysis to monitor for emergence of viral variants resistant to VX 787 and to oseltamivir | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (176):
- United States (129):
  - Athens, Alabama
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Huntsville, Alabama
  - Scottsboro, Alabama
  - Harrisburg, Arkansas
  - Phoenix, Arkansas
  - Anaheim, California
  - Burbank, California
  - Canoga Park, California
  - Chula Vista, California
  - El Cajon, California
  - Encino, California
  - Fresno, California
  - Garden Grove, California
  - Harbor City, California
  - Huntington Beach, California
  - La Mesa, California
  - Lomita, California
  - Long Beach, California
  - Norwalk, California
  - Oakland, California
  - Oceanside, California
  - Paramount, California
  - San Diego, California
  - Santa Monica, California
  - Tustin, California
  - Upland, California
  - Colorado Springs, Colorado
  - Northglenn, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Brooksville, Florida
  - Chiefland, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Doral, Florida
  - Edgewater, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Homestead, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Lake Worth, Florida
  - Lakeland, Florida
  - Long Beach Resort, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Anderson, Idaho
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Anderson, Indiana
  - Muncie, Indiana
  - Newburgh, Indiana
  - Council Bluffs, Iowa
  - Overland Park, Kansas
  - Bardstown, Kentucky
  - Hazard, Kentucky
  - Eunice, Louisiana
  - Mandeville, Louisiana
  - Shreveport, Louisiana
  - Oxon Hill, Maryland
  - Worcester, Massachusetts
  - Belton, Michigan
  - Niles, Michigan
  - Troy, Michigan
  - St Louis, Missouri
  - Fremont, Nebraska
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Rochester, New York
  - Rosedale, New York
  - Advance, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Morganton, North Carolina
  - Salisbury, North Carolina
  - Akron, Ohio
  - Dayton, Ohio
  - Hilliard, Ohio
  - Huber Heights, Ohio
  - Tulsa, Oklahoma
  - Harleysville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Warminster, Pennsylvania
  - East Providence, Rhode Island
  - Johnston, Rhode Island
  - Greer, South Carolina
  - Laurens, South Carolina
  - Mt. Pleasant, South Carolina
  - Rock Hill, South Carolina
  - Simpsonville, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Amarillo, Texas
  - Arlington, Texas
  - Austin, Texas
  - Baytown, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Humble, Texas
  - Katy, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Clinton, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Alexandria, Virginia
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (4):
  - Borgerhout
  - Linkebeek
  - Massemen
  - Wichelen
- Bulgaria (2):
  - Sofia
  - Veliko Tarnovo
- Canada (10):
  - Calgary, Alberta
  - West Vancouver, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - Brampton, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Mirabel, Quebec
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
  - Trois-Rivières, Quebec
- Estonia (5):
  - Paide
  - Saku
  - Tallinn
  - Tartu
  - Võru
- Germany (5):
  - Berlin
  - Essen
  - Goch
  - Hamburg
  - Stuhr
- Latvia (7):
  - Balvi
  - Daugavpils
  - Jelgava
  - Jēkabpils
  - Kuldīga
  - Lielvārde
  - Riga
- Toa Baja, Puerto Rico
- South Africa (13):
  - Boksburg
  - Breyten
  - Cape Town
  - Durban
  - Johannesburg
  - Kempton Park
  - Krugersdorp
  - Middelburg
  - Moloto South
  - Pretoria
  - Thabazimbi
  - Vanderbijlpark
  - Worcester

REFERENCES:
- [Derived] Finberg RW, Lanno R, Anderson D, Fleischhackl R, van Duijnhoven W, Kauffman RS, Kosoglou T, Vingerhoets J, Leopold L. Phase 2b Study of Pimodivir (JNJ-63623872) as Monotherapy or in Combination With Oseltamivir for Treatment of Acute Uncomplicated Seasonal Influenza A: TOPAZ Trial. J Infect Dis. 2019 Mar 15;219(7):1026-1034. doi: 10.1093/infdis/jiy547. PMID 30428049